CLINICAL TRIAL: NCT07049315
Title: Effect of Oral Mandibular Advancement Devices on Nocturnal Gastroesophageal Reflux in Adults With Obstructive Sleep Apnea: A Randomized Controlled Trial
Brief Title: Mandibular Advancement Devices for Reflux in Obstructive Sleep Apnea
Acronym: MAD-ROSA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tuiuti University of Paraná (Other)
Responsible Party: Principal Investigator, Flávio Magno Gonçalves, Professor, Tuiuti University of Paraná
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NEC01
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gastroesophageal reflux; Sleep Apnea, Obstructive
MeSH Terms: conditions — Gastroesophageal Reflux; Sleep Apnea, Obstructive | interventions — Occlusal Splints; Mandibular Advancement

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups:
  The experimental group will receive a mandibular advancement device (MAD) that repositions the lower jaw forward during sleep.
  The comparator group will receive a lower jaw oral device without mandibular advancement.
  Each participant will use the assigned device nightly for 6 months. There is no crossover between arms.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant, the primary investigator, and the assessor of outcomes will not know which device the participant receives. Only the provider who delivers the oral appliance will know.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandibular Advancement Device (MAD) (Experimental): Participants in this group will receive a custom-made mandibular advancement device (MAD), designed to reposition the lower jaw forward during sleep. The appliance is used nightly for 180 days and aims to improve upper airway patency and reduce nighttime gastroesophageal reflux episodes. The device is made of heat-cured acrylic and adjusted based on individual mandibular protrusion measurements.
  Interventions: Device: Mandibular Advancement Device
- Lower Oral Device Without Mandibular Advancement (DIO) (Active Comparator): Participants in this group will receive a lower jaw oral device that does not advance the mandible. The appliance is also indicated for patients with obstructive sleep apnea and provides dental disocclusion without altering jaw position. It will be used nightly for 180 days, serving as the control intervention. The device is fabricated similarly to the MAD but without mandibular repositioning.
  Interventions: Device: Lower Oral Device Without Mandibular Advancement

INTERVENTIONS:
Device: Mandibular Advancement Device — A custom-made intraoral appliance designed to reposition the mandible forward during sleep. The device increases the upper airway space by maintaining the lower jaw in a protruded position, aiming to reduce airway collapse and decrease nocturnal gastroesophageal reflux. It is fabricated from heat-cured acrylic based on individual dental impressions and bite registrations taken in a protruded mandibular position.
  Arms: Mandibular Advancement Device (MAD)
Device: Lower Oral Device Without Mandibular Advancement — A lower jaw oral appliance made of heat-cured acrylic, fabricated from standard dental impressions and bite registration in habitual occlusion. This device does not reposition the mandible but provides posterior dental disocclusion. It is also used in patients with obstructive sleep apnea and serves as an active comparator to evaluate the specific impact of mandibular advancement on nocturnal gastroesophageal reflux.
  Arms: Lower Oral Device Without Mandibular Advancement (DIO)

SUMMARY:
The purpose of this randomized clinical trial is to learn if a mandibular advancement device (a type of oral appliance) can help reduce nighttime acid reflux in adults with obstructive sleep apnea. The study also aims to understand whether this device can improve sleep quality and quality of life.

The main questions the study aims to answer are:

* Does using a mandibular advancement device reduce the number and intensity of nighttime reflux episodes?
* Does the device improve sleep and daily well-being in people with sleep apnea and reflux?

Researchers will compare two types of oral appliances:

* A mandibular advancement device, which moves the lower jaw forward during sleep
* A lower jaw oral device without advancement, which also aims to help people with sleep apnea but does not reposition the jaw

Participants will:

Wear the assigned oral device every night for 6 months Visit the clinic for check-ups and adjustments Complete short questionnaires about reflux symptoms, sleep quality, swallowing, diet, and quality of life Have saliva pH measured and X-rays taken before and after using the device This study hopes to find out whether oral devices can be a good option for people who do not tolerate CPAP therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years
* Clinical diagnosis of obstructive sleep apnea (OSA) confirmed by polysomnography type I
* Presence of nocturnal gastroesophageal reflux symptoms
* Not currently using CPAP therapy
* Dentate individuals able to wear oral devices
* Able and willing to comply with the study protocol
* Provided written informed consent

Exclusion Criteria:

* Severe OSA (Apnea-Hypopnea Index > 30)
* Current or recent use of proton pump inhibitors or other anti-reflux medications
* Neurological or neuromuscular disorders
* Use of removable dental prostheses (partial or total)
* Prior surgeries for apnea or reflux
* Known allergy or intolerance to dental acrylic materials
* Inability to attend follow-up visits or complete questionnaires

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in nocturnal gastroesophageal reflux symptoms using the N-GSSIQ questionnaire | Baseline and 180 days after intervention
  Participants will complete the Nocturnal Gastroesophageal Reflux Symptom Severity and Impact Questionnaire (N-GSSIQ), a validated scale ranging from 0 to 36, where higher scores indicate worse nocturnal reflux symptoms. Assessments will be performed at baseline and after 180 days of nightly oral device use to compare symptom severity between groups.

SECONDARY OUTCOMES:
Change in sleep quality using the Pittsburgh Sleep Quality Index (PSQI) | Baseline and 180 days after intervention
  The Pittsburgh Sleep Quality Index (PSQI), ranging from 0 to 21, where higher scores indicate worse sleep quality, will be administered at baseline and after 180 days of device use. The goal is to compare changes in global sleep quality scores between groups.
Change in daytime sleepiness using the Epworth Sleepiness Scale (ESS) | Baseline and 180 days after intervention
  The Epworth Sleepiness Scale (ESS), ranging from 0 to 24, where higher scores indicate greater daytime sleepiness, will be used to measure excessive sleepiness at baseline and after 180 days of using the assigned oral device. Scores will be compared between groups.
Change in salivary pH levels | Baseline and 180 days after intervention
  Salivary pH will be measured before and after the 180-day intervention period, using a standardized collection and digital pH meter. The goal is to assess whether the mandibular advancement device affects oral acidity associated with nocturnal reflux.
Change in quality of life using the WHOQOL-BREF questionnaire | Baseline and 180 days after intervention
  Participants will complete the World Health Organization Quality of Life - BREF (WHOQOL-BREF), which provides domain scores ranging from 0 to 100, where higher scores indicate better quality of life. Assessments will occur at baseline and after 180 days to compare changes between groups.

CONTACTS AND LOCATIONS:
Overall Officials: José Stechman-Neto, PhD, DDS, Study Director — Universidade Tuiuti do Paraná
Locations (1):
- Universidade Tuiuti do Paraná - Centro de Diagnóstico das Alterações Temporomandibulares (CDATM), Curitiba, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be made available upon reasonable request to the principal investigator, after primary results are published.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available starting in July 2027 and will remain accessible for 5 years (until July 2032).
Access Criteria: Qualified researchers with IRB/ethics committee approval